CLINICAL TRIAL: NCT07062978
Title: A Multicenter, Randomized, Double-blind Comparative Study to Valuating the Efficacy and Safety of QL1206 and Prolia® in Postmenopausal Women With Osteoporosis at High Risk of Fracture
Brief Title: A Comparative Study to Valuating the Efficacy and Safety of QL1206 and Prolia®
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL1206-305
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Postmenopausal Women With Osteoporosis at High Risk of Fracture
MeSH Terms: interventions — QL1206; Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1206 (Experimental): QL1206 Denosumab injection(60 mg)
  Interventions: Drug: QL1206
- Prolia® (Active Comparator): Prolia® Denosumab injection(60 mg)
  Interventions: Drug: Prolia®

INTERVENTIONS:
Drug: QL1206 — QL1206 Denosumab injection(60 mg) was administered subcutaneously once every 6 months for a maximum of 2 consecutive doses throughout the trial.
  Arms: QL1206
Drug: Prolia® — Prolia® Denosumab injection(60 mg) was administered subcutaneously once every 6 months for a maximum of 2 consecutive doses throughout the trial.
  Arms: Prolia®

SUMMARY:
This study is a multicenter, randomized, double-blind comparative study to valuating the efficacy and safety of QL1206 and Prolia® in postmenopausal women with osteoporosis at high risk of fracture.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who agree to participate in the study and sign the informed consent form.
* Postmenopausal women who can walk freely, aged 50-85 years (including 50 and 85 years old).
* Subjects whose absolute value of bone mineral density (BMD) in the lumbar or total hip area meets T values ≤ -2.5 and > -4.0.
* Subjects who must have at least one of the following risk factors: History of previous fragility fractures (occurring after the age of 40); history of hip fractures in fathers or mothers; increased bone turnover rate during screening; low body weight (BMI ≤ 19 kg/m2); advanced age (aged ≥ 65 years); current smoke.
* The duration of spontaneous amenorrhea was >2 years or >2 years after bilateral oophorectomy. If the status of bilateral oophorectomy is unknown or if the ovaries are preserved after hysterectomy, follicle stimulating hormone (FSH) levels >40mIU/mL may be used to confirm the status of postoperative menopause.

Exclusion Criteria:

* Bone/metabolic disease.
* Hyperparathyroidism or hypoparathyroidism.
* Thyroid condition: Hyperthyroidism or hypothyroidism.
* Rheumatoid arthritis.
* Malabsorption syndrome.
* Renal disease - severe impairment of kidney function.
* Vitamin D defViciency (25-hydroxyvitamin D, 25OHD <20 ng/mL).
* Oral or dental diseases: previous or current evidence of mandibular osteomyelitis or osteonecrosis; Acute dental or mandibular disease requiring oral surgery; Planning invasive dental surgery; Failure to recover from dental or oral surgery.
* Previously used denosumab drugs.
* Use of intravenous bisphosphonates, fluoride, or strontium to treat osteoporosis within the last 5 years.
* OOral bisphosphonates (used for at least 3 years, or used for less than 3 years but more than 3 months, with the last use occurring <1 year before the ICF).
* Use of any of the following drugs within 6 weeks prior to screening that may affect bone metabolism.
* History of more than two vertebral fractures.
* Malignant tumors.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in lumbar spine(LS)-BMD at Month 12 | Baseline and 12 months
  Percent Change From Baseline in lumbar spine(LS)-BMD at Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital Bijie Hospital, Guizhou, China